CLINICAL TRIAL: NCT04307719
Title: Carriers of Genetic Diseases in the Mexican Jewish Community
Brief Title: Prevalence of Carriers of Genetic Diseases in the Mexican Jewish Community
Status: Completed | Type: Observational
Sponsor: Anahuac University (Other)
Responsible Party: Principal Investigator, Dan Morgenstern-Kaplan, Principal Investigator, Anahuac University
Other Study IDs: 201944
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Genetic Predisposition; Carrier, Gestational
Keywords: Carrier Screening; Jewish
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Saliva samples for commercially available DNA carrier screening panels
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mexican Jewish Community: Sample of Patients from the Mexican Jewish Community to be subjected to genetic testing

SUMMARY:
The Jewish Population is at an increased risk for genetic diseases, especially autosomal recessive, thus, screening should be done to determine carrier status of several genetic diseases. In the Mexican Jewish Community, which is a very diverse community (regarding geographical origins), data of carrier status is unknown. The study aims to determine carrier prevalence for over 300 diseases using commercially available panels.

DETAILED DESCRIPTION:
Background: Preconceptional screening of genetic diseases is currently a underused and very useful tool, especially in populations that are at risk to be carriers of genetic diseases, such as the Jewish people, with carrier rates as high as 1:4 for any autosomal recessive disease. The Mexican Jewish Community is one of these populations at-risk, and there is no modern genetic research of the carrier rates in this community.

Goals: This research project in the Mexican Jewish Community aims to determine the prevalence of carriers in the community in order to properly generate in the future, a systematic carrier screening in the community.

Research Plan: The investigators propose a descriptive, observational, cross-sectional study, in which a representative sample of the Mexican Jewish Community (Which composes of Ashkenazi, Sephardic and Middle-Eastern Jews) of 250 patients, in which we´ll collect a saliva sample with a collection kit. Furthermore, the sample will be sent to a private commercial laboratory to perform the Comprehensive Carrier Screening to analyze the 301 genes included in the test plus the 13 add-on genes.

Analysis: Other demographic variables will be collected from the patients at the time of the sample collection to identify possible risk factors (geographical origin, number of Jewish grandparents, history of genetic diseases, et. al) and a correlation analysis will be performed to verify the strength of those risk factors on the carrier status of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Jewish Origin in at least 1 grandparent
* Members of one of the Jewish sub-Communities in Mexico City

Exclusion Criteria:

* Pregnant Women

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Representative sample of the Mexican Jewish Community of child-bearing age, of both sexes.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Carrier Status for 300+ Genetic Diseases | 30 days after sample collection
  Patients will be screened for over 300 genetic diseases to determine carrier status

CONTACTS AND LOCATIONS:
Overall Officials: Dan Morgenstern-Kaplan, MD, Principal Investigator — Anahuac University
Locations (1):
- Universidad Anáhuac México, Huixquilucan, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: No